CLINICAL TRIAL: NCT05316870
Title: Construction and Evaluation of Standardized Anticoagulant Management Model of Atrial Fibrillation in Primary Medical Institutions Under Hierarchical Diagnosis and Treatment System
Brief Title: Construction and Effect Evaluation of Anticoagulation Management Model in Atrial Fibrillation
Acronym: AMS-AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Municipal Health Commission (Other Government)
Collaborators: Exhibition Road Community Health Service Center of Xicheng District, Beijing, China (Unknown); Xinjiekou Community Health Service Center of Xicheng District, Beijing, China (Unknown); Guanwai Community Health Service Center of Xicheng District, Beijing, China (Unknown); Guannei Community Health Service Center of Xicheng District, Beijing, China (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CFH 2020-4-7025
Record Dates: First submitted 2022-01-25; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Anticoagulation management plan and process; Primary medical institutions
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Each community health service center randomly included patients with atrial fibrillation who met the admission criteria into the trial group or the control group. The intervention measures are the standardized anticoagulation management plan and process of atrial fibrillation in primary medical institutions.
Who Masked: Participant
Masking Description: Single Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The standardized anticoagulation management program of atrial fibrillation in primary medical institutions was implemented for the patients with atrial fibrillation in the intervention group.
  Interventions: Behavioral: Standardized anticoagulation management plan and process of atrial fibrillation in primary medical institutions
- Control group (Other): The current general practitioner management mode was continued for the patients with atrial fibrillation in the control group.
  Interventions: Behavioral: Conventional general practitioner management model

INTERVENTIONS:
Behavioral: Standardized anticoagulation management plan and process of atrial fibrillation in primary medical institutions — Compared with the current anticoagulation management service, we pay more attention to early initiation of anticoagulant therapy and long-term follow-up management.
  Arms: Intervention group
Behavioral: Conventional general practitioner management model — The current general practitioner anticoagulation management model was continued in the control group.
  Arms: Control group

SUMMARY:
Study types and hypotheses: multicenter randomized controlled trials. This study predicts that standardized anticoagulation management of atrial fibrillation in primary health care institutions can reduce the prevalence of atrial fibrillation stroke by 50%.

1. Formulation and revision of standardized anticoagulation management plan and process for atrial fibrillation in primary health care institutions.

   Using the mature anticoagulation management model of atrial fibrillation for reference, based on the clinical data and disease management needs of patients with atrial fibrillation in five community health service centers in Xicheng District of Beijing. To formulate the anticoagulation management plan and process of atrial fibrillation suitable for grass-roots medical institutions. After the completion of the first draft of anticoagulation management plan and process, two rounds of multi-disciplinary experts were organized to demonstrate the feasibility and scientific nature of the first draft. Finally, based on the practice and effect evaluation of clinical application management, the scheme is revised and improved.
2. To evaluate the feasibility and clinical application effect of standardized anticoagulation management scheme and process for atrial fibrillation.

First of all, the baseline clinical database of patients with multicenter atrial fibrillation was established; secondly, patients with atrial fibrillation who met the entry criteria were randomly included in the trial group or control group and followed up for two years. The anticoagulation treatment rate, the incidence of bleeding and thromboembolic events, anticoagulation compliance rate and knowledge awareness rate of atrial fibrillation in the two groups were compared, and the effect of standardized anticoagulation management of atrial fibrillation in primary medical institutions was evaluated.

DETAILED DESCRIPTION:
To organize experts to formulate a standardized anticoagulation management plan and process for atrial fibrillation in grass-roots medical institutions

1. Write the first draft of "standardized anticoagulation management plan and process of atrial fibrillation in primary medical institutions" By searching the anticoagulation management guidelines and expert consensus of atrial fibrillation at home and abroad, do a comparative study, determine the main points of anticoagulation management; analyzing the baseline clinical database of patients with multicenter atrial fibrillation, combined with quantitative and qualitative research, to explore the anticoagulation management needs of patients with atrial fibrillation. Based on the above results, the first draft of standardized anticoagulation management plan and process of atrial fibrillation in grass-roots medical institutions was written.
2. Organize expert group interviews. A multidisciplinary expert group was identified, including cardiology, neurology, general medicine, nursing and pharmacy, with 1 or 2 middle-level and above professionals selected in each discipline. Design the interview outline, according to the interview outline, a senior general practitioner encourages and guides the team members to express their own views on the subject. The main contents include: how scientific is this anticoagulation management scheme? What is the value of clinical application? What are the difficulties in the implementation process? What are the contents that need to be further improved?
3. Revision and improvement of "standardized anticoagulation management scheme and process for atrial fibrillation in primary medical institutions" According to the results of the expert group interview, revise and further improve the "standardized anticoagulation management plan and process of atrial fibrillation in primary medical institutions" to generate the final intervention plan.

To evaluate the clinical effect of standardized anticoagulation management scheme and process for atrial fibrillation.

1. Observation indicators Main outcome measures: the rate of anticoagulant therapy, the rate of reaching the standard of INR, the incidence of bleeding and thromboembolic events at 3 months, 6 months, 9 months, 12 months, 18 months and 24 months.

   Secondary indicators: anticoagulant compliance rate and knowledge awareness rate of atrial fibrillation at 6 months, 12 months and 18 months. Blood routine: hemoglobin, platelet; biochemistry: glutamic pyruvic transaminase, glutamic oxaloacetic transaminase, serum creatinine, urea nitrogen, glomerular filtration rate; electrocardiogram / dynamic electrocardiogram, echocardiography.
2. Follow-up plan Patients' symptoms and signs, diet and exercise in the process of anticoagulation management were followed up once a month, and when unmanageable new symptoms or drug side effects appeared, they were referred to secondary or tertiary hospitals for treatment in time; a regular comprehensive physical examination was arranged once a year, including blood routine, biochemical, ECG / dynamic electrocardiogram, echocardiography, etc., and the follow-up period was 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old, regardless of sex.
* It is consistent with the diagnostic basis of atrial fibrillation in "Atrial Fibrillation: current Cognition and treatment recommendations-2018".
* Receive oral anticoagulant therapy, such as warfarin or NOACs, as needed.
* There is a contracted family doctor (if not, they can be included in the study after guiding them to sign up for a family doctor).
* Have certain reading comprehension ability, be able to follow up regularly, have good compliance, and select the residents living in the vicinity.
* Volunteer to participate in this clinical study and sign a written informed consent form

Exclusion Criteria:

* Other diseases requiring anticoagulant therapy, such as pulmonary embolism, were included in the group.
* Suffer from severe mental illness or serious diseases that affect their survival, such as AIDS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2020-09-04 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Anticoagulant treatment rate, % | Change from Baseline Anticoagulant treatment rate at 24 months
  Anticoagulant therapy rate (%) = number of people actually receiving anticoagulant therapy / number of people who should receive anticoagulant therapy x 100%anticoagulant therapy / the total number of people who should receive anticoagulant therapy x 100%.
Incidence of bleeding and thromboembolic events | Change from Baseline bleeding and thromboembolic events rate at 24 months
  Incidence of thromboembolic events / anticoagulation related bleeding events (%) = number of thromboembolic events / anticoagulation related bleeding events in a certain period / number of people observed in the same period x 100% (unit: person year)
INR compliance rate | Change from 12 months INR compliance rate at 24 months
  INR compliance rate (%) = the number of INR compliance (2.0 / 3.0) / the total number of INR monitored in the same period × 100%

SECONDARY OUTCOMES:
Anticoagulant compliance rate | Change from 12 months INR compliance rate at 24 months
  Using the Chinese revised version of Morisky Drug Compliance scale
Knowledge awareness rate of atrial fibrillation | Change from 12 months INR compliance rate at 24 months
  Awareness rate = the number of correct questions answered by the respondents / the total number of questions answered by the respondents x 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Xia J Wang, Master, Study Chair — FuXing Hospital, Capital Medical University
Locations (1):
- Yuetan Community Health Service Center Fu Xing Hospital, Capital Medical University, Beijing, Beijing Municipality, China